CLINICAL TRIAL: NCT03718650
Title: Total Tumor Mapping (TTM) for Resectable Pancreatic Cancer: Establishing the Radiomic/Pathologic Foundation of Heterogeneity
Brief Title: Total Tumor Mapping (TTM) for Resectable Pancreatic Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-19599
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Cancer; Resectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pimonidazole; Pancreaticoduodenectomy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Scans, Surgical Resection and Assessment (Experimental): Pre-surgery scans, surgical resection and post-surgery pathological assessment. All patients will receive standard of care imaging and blood tests. If suitable, non-standard of care abdominal MRI imaging will be done. 16-24 hours prior to surgery, patients will be administered a single dose of 0.5 g/m^2 pimonidazole (HydroxyProbe).
  Interventions: Drug: Pimonidazole; Procedure: Surgical Resection

INTERVENTIONS:
Drug: Pimonidazole — Patients will take a single dose of 0.5 g/m^2 (approximately 13 mg/kg) of oral pimonidazole HCI 16 to 24 hours prior to surgery.
  Other Names: HydroxyProbe; Pimonidazole HCI
Procedure: Surgical Resection — Patients will undergo Pancreaticoduodenectomy or Whipple procedure, which involves the resection of the pancreatic head, duodenum, gallbladder, and a portion of the stomach, 16 to 24 hours after consuming oral pimonidazole.
  Other Names: Whipple Procedure; Pancreatoduodenectomy; Surgery

SUMMARY:
At present there is no validated prognostic tool for patients with resectable pancreatic cancer (RPC) to determine how best to tailor individual therapy. This study is to see if tumor features in blood and imaging prior to surgery correspond with tumor heterogeneity in the specimen after surgery.

DETAILED DESCRIPTION:
This study is to prospectively determine whether there is a predictive relationship in RPC between pre-operative radiomic imaging features and pathologic tumor heterogeneity, delineated by gene-expression-based RSI and histologic measures of hypoxia measured by Glut-1 and CA-IX as well as the degree of pimonidazole staining.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older who have biopsy-proven resectable pancreatic cancer
* Participants must have a histological diagnosis of pancreatic head ductal adenocarcinoma at least ≥ 1 cm from ampula.
* Participants must be able to undergo all 3 imaging modalities.
* Participants' medical statuses must be considered appropriate for surgery and for general anesthesia.
* Female participants and female partners of male participants undergoing optional PET-CT or CT pancreatic protocol scan cannot be pregnant or nursing, as confirmed by serum pregnancy test if the patient is a woman of child-bearing potential.
* All female participants of child-bearing potential must agree to use birth control, including oral, injectable, or mechanical contraception, abstinence, or vasectomy for 30 days following pimonidazole administration.
* Adequate kidney and liver function as assessed by laboratory studies. Laboratory studies must be completed within 28 days prior to pimonidazole administration;
* Must be capable of providing informed consent and demonstrate a willingness to comply with all the study procedures and visits;
* Must be able to undergo MRI scans without having a pacemaker or other indwelling metal, which would contraindicate the scan.
* Have an Eastern Cooperative Oncology Group (ECOG) score of 0 to 2.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Participants who are contraindicated for MRI or gadolinium contrast agents.
* If the patient has an iodine contrast allergy, they must be able to take standard pre-medications so they can safely undergo a CT scan.
* Participants with a known active cancer with a prognosis that would contraindicate a curative intent pancreatic resection.
* Participants with depressed liver function, as assessed with a screening liver function test yielding serum ALT or AST greater than the IULN or total bilirubin greater than 2 mg/dL.
* Presence of any other co-existing condition, which, in the judgment of the investigator, might increase the risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Radiosensitivity Index and Degree of Pimonidazole Staining | Up to 14 weeks
  Relationship between PET/CT, MRI or pancreas protocol CT features and the pathological correlations of radiation sensitivity and hypoxia, as measured by the radiosensitivity index (RSI) and degree of pimonidazole staining in resectable pancreatic cancer.

SECONDARY OUTCOMES:
Correlative Biomarkers | Up to 14 weeks
  Investigators will quantitiatively compare correlative biomarkers with the degree of pimonidazole staining and RSI. These biomarkers will include radiomic features from the preoperative imaging tests, serum CA 19-9, and histological markers for biological hypoxia, GLUT-1, and CA-IX. Data from all of these biomarkers will be available as continuous variables. The association between RSI (or % pimonidazole-positive pixels) and biomarkers will be assessed using the Spearman correlation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hoffe, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States